CLINICAL TRIAL: NCT05121103
Title: A Phase 1/1b, Open-label Multi-center Two-part Study of SETD2 Inhibitor EZM0414 in Subjects With Relapsed/Refractory Multiple Myeloma and Relapsed/Refractory Diffuse Large B Cell Lymphoma
Brief Title: A Study of the Safety, Tolerability and Effectiveness of EZM0414 (IPN60210) Investigative Product in Participants With Relapsed/Refractory Multiple Myeloma and Relapsed/Refractory Diffuse Large B Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic business decision
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SET-101
Record Dates: First submitted 2021-10-18; First posted 2021-11-16 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma, Refractory; Diffuse Large B-Cell Lymphoma; Diffuse Large B Cell Lymphoma Refractory; Multiple Myeloma in Relapse
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label EZM0414 (Experimental): Participants will receive EZM0414 in continuous 28-day cycles. EZM0414 will be administered orally once daily (QD) without food.
  Participants who receive EZM0414 at Maximum tolerated dose (MTD) and do not have Dose limiting toxicities (DLT) in the dose escalation part of the study will be rolled over to a cohort of this dose expansion part.
  Cohort 1 for R/R MM Participants. Cohort 2 for R/R MM Participants. Cohort 3 for Participants with R/R DLBCL.
  Interventions: Drug: EZM0414

INTERVENTIONS:
Drug: EZM0414 — Immediate-release film-coated tablets: Six dose levels starting at 100 mg, and then 200 mg, 300 mg, 400 mg, 600 mg, and 900 mg as well as an optional step-down dose level of 75 mg (if needed)
  Other Names: IPN60210

SUMMARY:
This study will include participants with relapsed/refractory (R/R) Multiple Myeloma (MM). MM is a type of cancer of the blood. This study will also include participants with relapsed/refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL).

DLBCL is also a type of cancer of the blood. They are referred to as 'relapsed' when the disease has come back after treatment and 'refractory' when treatment no longer works. The study has 2 main parts, called phase 1 and phase 1b. The main objective of both parts will be to evaluate the safety and tolerability of the study drug, called EZM0414.

The main objective of phase 1b will also be to determine the effectiveness of EZM0414. During phase 1 six dose levels will be tested to obtain the most tolerated dose. Participants will receive study drug at the assigned dose level every 28 days. During phase 1b participants will receive study drug at the maximum tolerated dose in 28-day cycles.

DETAILED DESCRIPTION:
The first part of the study will be a Phase 1 dose-escalation designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of EZM0414 in subjects with R/R MM and R/R DLBCL.

Six dose levels starting at 100 mg, then 200 mg, 300 mg, 400 mg, 600 mg, and 900 mg as well as an optional step-down dose of 75 mg (if needed) will be tested. The second part of the study is the Phase 1b dose expansion at the MTD designed to evaluate safety and efficacy in subjects with R/R DLBCL and R/R MM with or without select genetic translocation.

Dose expansion will enroll subjects in 3 cohorts: Cohort 1 for R/R MM subjects with t(4;14), Cohort 2 for R/R MM subjects without t(4;14), and Cohort 3 for subjects with R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide signed informed consent after review of verbal and written material about the trial and agree to abide with protocol requirements. All study related activities must be carried out after written consent is obtained.
2. Subjects must be ≥18 years of age at the time of signing the ICF (Informed Consent Form).
3. Subjects must have an Eastern Cooperative Oncology Group (ECOG) status of 0 - 2.
4. For MM, subjects must have measurable disease by IMWG (International Myeloma Working Group) 2016 criteria
5. For DLBCL, subjects must have measurable disease by Lugano criteria
6. Females must not be breastfeeding or pregnant at screening
7. Females of childbearing potential must not have had unprotected sexual intercourse while participating in this study
8. Male subjects must either practice complete abstinence or agree to use a latex or synthetic condom, even with a successful vasectomy, during study treatment and for 30 days after the final dose of study treatment

Exclusion Criteria:

1. Subjects with plasma cell leukemia defined as a plasma cell count >2000/mm3.
2. Subjects with Waldenstrom's macroglobulinemia or smoldering MM.
3. Subjects who had prior treatment with SETD2 or NSD2 inhibitor.
4. Subjects with active acute or chronic systemic infection requiring systemic treatment, including COVID-19.
5. Has cardiovascular impairment
6. Prolongation of corrected QT interval using Fridericia's formula (QTcF) to > 480 msec or history of long QT syndrome.
7. Known left ventricular ejection fraction (LVEF) < 50% by either echocardiogram (ECHO) or multigated acquisition (MUGA).
8. Prior major surgery within 4 weeks of treatment start.
9. Known hypersensitivity to components of the investigational product.
10. Subjects who have received treatment with any unapproved drug product within 4 weeks prior to screening.
11. Current participation in any other interventional clinical study except for follow up.
12. Subjects with a history of or active malignancy other than disease under study
13. Underlying medical/social conditions that in PI opinion will place the subject in significant risk and affect the interpretation of toxicity and adverse events assessments.
14. Inability to take oral medication or known gastrointestinal (GI) disease, GI procedure or medical condition that could interfere with the oral absorption or tolerance of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Astera Cancer Care, East Brunswick, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Baylor University Medical Center (Texas Oncology), Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2025/05/05090658/set-101-Lay-Results-Synopsis-English_29-Apr-2025.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This first-in-human, Phase I/Ib, open-label, multi-center study was conducted in participants with relapsed/refractory (R/R) multiple myeloma (MM) and R/R diffuse large B cell lymphoma (DLBCL) at 15 investigational sites for Part 1 (dose escalation). The study was planned to be conducted in 2 parts: Part 1 and Part 2 (dose expansion). The study was terminated prior to completing Part 1 of the study. Part 2 was not started.
Pre-assignment Details: The study was planned to have a screening period (28 days), treatment period (Part 1 and Part 2) and safety follow-up period (30 days). Due to early study termination, only results of the Part 1 are presented. A total of 13 participants were enrolled in Part 1 of the study. EZM0414 is also referred to as IPN60210.
Groups:
- Part 1: EZM0414 100 mg: Participants with translocation (t)(4;14) R/R MM or non-t(4;14) R/R MM or R/R DLBCL received EZM0414 100 milligrams (mg) tablet orally once daily (QD) in continuous 28-day cycles (except on Days 2 and 3 of Cycle 1) until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
- Part 1: EZM0414 200 mg: Participants with t(4;14) R/R MM or non-t(4;14) R/R MM or R/R DLBCL received EZM0414 200 mg tablet orally QD in continuous 28-day cycles (except on Days 2 and 3 of Cycle 1) until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
- Part 1: EZM0414 300 mg: Participants with t(4;14) R/R MM or non-t(4;14) R/R MM or R/R DLBCL received EZM0414 300 mg tablet orally QD in continuous 28-day cycles (except on Days 2 and 3 of Cycle 1) until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
Period: Overall Study
Arm/Group | Part 1: EZM0414 100 mg | Part 1: EZM0414 200 mg | Part 1: EZM0414 300 mg
Started | 4 | 3 | 6
Completed | 0 | 0 | 0
Not Completed | 4 | 3 | 6
Not completed — Progressive disease | 2 | 1 | 6
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of the study treatment in Part 1.
Groups:
- Part 1: EZM0414 100 mg: Participants with t(4;14) R/R MM or non-t(4;14) R/R MM or R/R DLBCL received EZM0414 100 mg tablet orally QD in continuous 28-day cycles (except on Days 2 and 3 of Cycle 1) until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
- Total: Total of all reporting groups
Arm/Group | Part 1: EZM0414 100 mg | Part 1: EZM0414 200 mg | Part 1: EZM0414 300 mg | Total
Number analyzed (Participants) | 4 | 3 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (7.42) | 70.3 (6.66) | 68.0 (13.11) | 66.5 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 8
  Male | 2 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 2 | 5 | 10
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 1 | 2 | 3 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event was any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product and which does not necessarily had a causal relationship with this treatment. A serious adverse event was any untoward medical occurrence that at any dose, resulted in death, was life-threatening, required in-subject hospitalization or prolongation of hospitalization, resulted in persistent or significant disability or incapacity, or resulted in a congenital abnormality or birth defect, was an important medical event. A TEAE was an AE that started or worsened in severity on or after the date of the first dose of the study treatment through 30 days after the end of treatment.
Time Frame: From first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment (Day 57), up to approximately 87 days
Population: The safety population included all participants who received at least 1 dose of the study treatment in Part 1. The study was terminated prior to completing Part 1 of the study. Part 2 was not started.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: EZM0414 100 mg | Part 1: EZM0414 200 mg | Part 1: EZM0414 300 mg
Number analyzed (Participants) | 4 | 3 | 6
Participants
  TEAEs | 3 | 3 | 6
  TESAEs | 1 | 0 | 1

2. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: According to National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0, DLT was defined as any of following AE that occurred in Part 1 during first cycle of study treatment: grade (G)4 neutropenia lasting >5 days; G3 febrile neutropenia; G3 thrombocytopenia with clinically significant bleeding; G4 thrombocytopenia; G4 anemia unexplained by underlying disease; any other non-hematological toxicity ≥3 except: alopecia, G3 nausea/vomiting or diarrhea for <3 days with supportive care, G3 fatigue for <1 week, G3 or higher isolated electrolyte abnormalities for up to 3 days, not clinically complicated, and resolved spontaneously, or responded to conventional medical interventions; G3 or higher amylase/lipase elevation without symptoms of pancreatitis; G3 tumor lysis syndrome for up to 3 days, not clinically complicated, and resolved spontaneously, or responded to conventional medical interventions; and any participant meeting Hy's law criteria.
Time Frame: From first dose of study treatment (Cycle 1 Day 1) up to end of the Cycle 1 (Cycle 1 Day 28), maximum of 28 days
Population: The DLT evaluable population included dose escalation dose level participants in the Safety population who received at least 80% of planned study treatment during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: EZM0414 100 mg | Part 1: EZM0414 200 mg | Part 1: EZM0414 300 mg
Number analyzed (Participants) | 4 | 3 | 6
Participants | 0 | 0 | 0

3. Primary Outcome: Part 2: Objective Response Rate (ORR)
Description: ORR was planned to be assessed in Part 2. ORR was defined as percentage of responders as assessed by Investigator per International Myeloma Working Group (IMWG) 2016 guidelines for MM (complete response [CR], stringent CR [sCR], partial response [PR], very good PR [VGPR]) or Lugano 2014 guidelines for DLBCL (CR+PR). Per IMWG response criteria, CR: negative immunofixation on serum and urine; disappearance of soft tissue plasmacytomas; <5% plasma cells in bone marrow(BM); sCR: CR + normal free light chain (FLC) ratio; absence of BM clonal cells by immunohistochemistry; VGPR: serum and urine M-protein (MP) detected by immunofixation but not on electrophoresis or ≥90% reduction in serum MP + urine MP<100 mg/24 hours (h) or ≥90% decrease in sum of maximal perpendicular diameter (SPD) compared to baseline in soft tissue plasmacytoma; PR: ≥50% reduction of serum MP and reduction in 24 h urinary M-protein by ≥90% or to <200 mg/24 h; ≥50% reduction in size (SPD) of soft tissue plasmacytomas.
Time Frame: Tumour assessments were planned to be performed at Screening (within 28 days before start of study treatment) or Cycle 1 Day 1 (pre-dose) up to end of the study, approximately 23 months
Population: The study was terminated prior to completing Part 1 of the study. Part 2 was not started.
Groups:
- Part 2: Cohort 1: R/R MM With t(4;14): Participants with R/R MM with t(4;14) were planned to receive EZM0414 tablet at maximum tolerated dose (MTD) orally QD in continuous 28-day cycles until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
- Part 2: Cohort 2: R/R MM Without t(4;14): Participants with R/R MM without t(4;14) were planned to receive EZM0414 tablet at MTD orally QD in continuous 28-day cycles until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
- Part 2: Cohort 3: R/R DLBCL: Participants with R/R DLBCL were planned to receive EZM0414 tablet at MTD orally QD in continuous 28-day cycles until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
Arm/Group | Part 2: Cohort 1: R/R MM With t(4;14) | Part 2: Cohort 2: R/R MM Without t(4;14) | Part 2: Cohort 3: R/R DLBCL
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Part 2: Progression-free Survival (PFS)
Description: PFS was planned to be assessed in Part 2. PFS was defined as the time from start of treatment until the first documented progressive disease (PD), as assessed by Investigator per IMWG 2016 guidelines for MM or Lugano 2014 guidelines for DLBCL or death due to any cause, whichever occurred first. Per IMWG response criteria, PD was defined as any 1 or more of the following criteria: a) increase of ≥25% from lowest confirmed value in either serum MP, serum MP increase ≥1 gram/deciliter (g/dL) if the lowest M-component was ≥5 g/dL or urine M-component, b) appearance of new lesion(s), ≥50% increase from nadir in SPD of >1 lesion, or ≥50% increase in the longest diameter of a previous lesion >1 centimeter (cm) in short axis.
Time Frame: as for outcome 3
Population: The study was terminated prior to completing Part 1 of the study. Part 2 was not started.
Groups:
- Part 2: Cohort 1: R/R MM With t(4;14): Participants with R/R MM with t(4;14) were planned to receive EZM0414 tablet at MTD orally QD in continuous 28-day cycles until consent withdrawal, unacceptable toxicity, disease progression or need for treatment prohibited on this study.
Arm/Group | Part 2: Cohort 1: R/R MM With t(4;14) | Part 2: Cohort 2: R/R MM Without t(4;14) | Part 2: Cohort 3: R/R DLBCL
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Part 2: Disease Control Rate (DCR)
Description: DCR was planned to be assessed in Part 2.DCR was defined as percentage of participants with confirmed CR,sCR,PR,VGPR,minimal response(MR) or stable disease(SD) per IMWG 2016 guidelines for MM/CR,PR, or SD per Lugano 2014 guidelines for DLBCL.Per IMWG response criteria,CR:negative immunofixation on serum and urine;disappearance of soft tissue plasmacytomas;<5% plasma cells in BM; sCR:CR+normal FLC ratio;absence of BM clonal cells by immunohistochemistry; VGPR:serum and urine MP detected by immunofixation but not electrophoresis or ≥90% reduction in serum MP+urine MP<100 mg/24h or ≥90% decrease in SPD in soft tissue plasmacytoma; PR:≥50% reduction of serum MP and reduction in 24h urinary M-protein by ≥90% or to <200mg/24h;≥50% reduction in size(SPD) of soft tissue plasmacytomas. MR:≥25% but ≤49% reduction in serum MP and reduction in 24h urine MP by 50-89%, which exceed 200 mg/24h; ≥50% reduction in size(SPD) of soft tissue plasmacytomas.SD:Not meeting criteria for CR,VGPR,PR,MR, or PD.
Time Frame: as for outcome 3
Population: The study was terminated prior to completing Part 1 of the study. Part 2 was not started.
Arm/Group | Part 2: Cohort 1: R/R MM With t(4;14) | Part 2: Cohort 2: R/R MM Without t(4;14) | Part 2: Cohort 3: R/R DLBCL
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Part 2: Duration of Response (DOR)
Description: DOR was planned to be assessed in Part 2. DOR was defined as the time from initial CR or PR to documented progression or death, whichever came first, as assessed by Investigator per IMWG 2016 guidelines for MM or Lugano 2014 guidelines for DLBCL. Per IMWG response criteria, CR: negative immunofixation on serum and urine; disappearance of any soft tissue plasmacytomas; <5% plasma cells in BM. PR: ≥50% reduction of serum MP and reduction in 24 h urinary M-protein by ≥90% or to <200 mg/24 h; ≥50% reduction in the size (SPD) of soft tissue plasmacytomas. PD: any 1 or more of the following criteria: a) increase of ≥25% from lowest confirmed value in either serum MP, serum MP increase ≥1 g/dL if the lowest M-component was ≥5 g/dL or urine M-component, b) appearance of new lesion(s), ≥50% increase from nadir in SPD of >1 lesion, or ≥50% increase in the longest diameter of a previous lesion >1 cm in short axis.
Time Frame: as for outcome 3
Population: The study was terminated prior to completing Part 1 of the study. Part 2 was not started.
Arm/Group | Part 2: Cohort 1: R/R MM With t(4;14) | Part 2: Cohort 2: R/R MM Without t(4;14) | Part 2: Cohort 3: R/R DLBCL
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment (Day 57), up to approximately 87 days. All-cause mortality (death) was assessed from first dose of study treatment (Day 1) up to early termination of the study, approximately 23 months.
Description: The safety population included all participants who received at least 1 dose of the study treatment in Part 1. The study was terminated prior to completing Part 1 of the study. Part 2 was not started.
Arm/Group | Part 1: EZM0414 100 mg | Part 1: EZM0414 200 mg | Part 1: EZM0414 300 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: EZM0414 100 mg (N=4) | Part 1: EZM0414 200 mg (N=3) | Part 1: EZM0414 300 mg (N=6)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: EZM0414 100 mg (N=4) | Part 1: EZM0414 200 mg (N=3) | Part 1: EZM0414 300 mg (N=6)
Platelet count decreased (Investigations) | 1 (1) | 2 (4) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (4) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (4)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated prior to completing Part 1 due to business reasons. Study termination was not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT05121103/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT05121103/SAP_001.pdf